CLINICAL TRIAL: NCT03419000
Title: Circulating microRNAs as Biomarkers of RESPIratory Dysfunction in Patients With Refractory epilePSY
Acronym: MIRESPILEPSY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL17_0666; 2017-A03307-46 (Other: ID-RCB)
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2022-04

CONDITIONS: Drug Resistant Epilepsy
Keywords: GTCS; Epilepsies, Partial; Drug Resistant Epilepsy; Circulating MicroRNA; Diagnostic
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsies, Partial; Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient (Experimental): Patients suffering from drug-resistant focal epilepsy or from drug-resistant generalized epilepsy according to ILAE classification and undergoing long-term video-EEG monitoring in Epilepsy unit of Lyon to record and characterize her/his seizure
  Interventions: Genetic: blood sample
- healthy volunteers (Active Comparator): Adult (≥ 18 years) Without history of neurological disorders and/or psychiatric disorders, and/or general medical disorders
  Interventions: Genetic: blood sample

INTERVENTIONS:
Genetic: blood sample — Seven blood samples (4 ml each on 5 EDTA and 2 dry tubes) will be collected in each patient/ healthy volunteers subject to determine the expression profile of miRNAs in the plasma as well as in the exosomes

SUMMARY:
Sudden and unexpected death in epilepsy (SUDEP) has become a major issue for patients with epilepsy and their physicians. SUDEP is a nontraumatic and non-drowning death in patients with epilepsy, unrelated to a documented status epilepticus, in which postmortem examination does not reveal a toxicologic or anatomic cause of death. It primarily affects young adults with drug-resistant epilepsy, with an incidence of about 0.5%/year. A recent study reported that up to 20% of patients with childhood onset drug resistant epilepsy will die of a SUDEP by the age of 45. Apart from optimizing antiepileptic drugs, no preventive treatment is available to prevent SUDEP. As underscored by the World Health Organization (WHO), there is an urgent need to develop specific therapeutic approaches to tackle this issue.

The primary objective of the proposal is to evaluate the diagnostic value of a set of circulating microRNAs pre-selected because of their implication in the regulation of molecular pathways involved in the respiratory regulation to identify patients with seizure-related respiratory dysfunction, as defined by occurrence ictal/peri-ictal pulse oxymetry < 90%.

A total of 50 patients will be included over a period of one year. Patients undergoing long-term video-EEG/SEEG monitoring will be recruited in the epilepsy monitoring unit of the Department of Functional Neurology and Epileptology, Hospices Civils de Lyon, Lyon, France.

It will be a case-control study in a cohort of patients with drug-resistant focal epilepsy undergoing long-term video-EEG monitoring, in which patients who demonstrate ictal/post-ictal hypoxemia (cases) will be compared with those without seizure-related respiratory dysfunction (controls).

ELIGIBILITY:
Inclusion Criteria:

For the patients :

* Adult patient (≥ 18 years) suffering from drug-resistant focal epilepsy or from drug-resistant generalized epilepsy according to ILAE classification
* Patient undergoing long-term video-EEG monitoring in Epilepsy unit of Lyon to record and characterize her/his seizure
* Patient who gave her/his written informed consent to participate to the study
* Patient affiliated to the French health care system

For the healthy volunteers :

* Adult (≥ 18 years)
* Without history of neurological disorders and/or psychiatric disorders, and/or general medical disorders
* Subject who gave her/his written informed consent to participate to the study
* Subject affiliated to the French health care system

Exclusion Criteria:

For the patients :

* Ongoing major depressive episode as defined by a score ≥ 15 at the French version of the NDDI-E scale*
* Current panic disorder as defined by a score ≥ 7 at the French version of the GAD-7 scale*
* Ongoing treatment with selective serotonin reuptake inhibitor
* Patient who benefit from a protective measure

For the healthy volunteers :

* Presence of the symptoms of anxiety and/or depression as defined by a score ≥ 11 at the French version of the Hospital Anxiety and Depression Scale (HADS)
* Ongoing treatment with selective serotonin reuptake inhibitor
* Subjects with these psychiatric comorbidities and/or treatment will be excluded in order to limit risk that the relation previously reported between miR-135a, miR-16, miR-1202 and depression and/or panic disorder and/or response to selective serotonin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Relation between the expression level of circulating microRNAs and the occurrence of SpO2 <90% during at least 5 seconds within the course of the seizure and/or within the five minutes following the end of the seizure | Day 0
  The primary objective of the proposal is to evaluate the diagnostic value of a set of circulating microRNAs pre-selected because of their implication in the regulation of molecular pathways involved in the respiratory regulation to identify patients with seizure-related respiratory dysfunction, as defined by occurrence ictal/peri-ictal pulse oxymetry < 90%

SECONDARY OUTCOMES:
Relation between the expression level of circulating microRNAs and the desaturation nadir | Day 0
  Evaluating the relation between a set of circulating microRNAs and the severity of the seizure-related respiratory dysfunction, as defined by the desaturation nadir
Relation between the expression level of circulating microRNAs and the patient's age | Day 0
Relation between the expression level of circulating microRNAs and the epilepsy duration | Day 0
Relation between the expression level of circulating microRNAs and the total number of seizures (ie focal seizures and GTCS) over the past three months | Day 0
Relation between the expression level of circulating microRNAs and the Number of GTCS over the past three months | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain RHEIMS, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Hospices Civils de Lyon, Bron
  - Service de Neurophysiologie Clinique Hôpital La Timone, Marseille